CLINICAL TRIAL: NCT00002328
Title: Oral/Intravenous Azithromycin in the Treatment of Cryptosporidiosis in Patients Whose Disease Has Not Been Controlled by Conventional Therapy
Brief Title: Azithromycin in the Treatment of Cryptosporidiosis in Patients Who Have Not Had Success With Other Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 058J; 066-167S
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Antidiarrheals; Cryptosporidiosis; Diarrhea; Acquired Immunodeficiency Syndrome; Azithromycin
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; Diarrhea; Acquired Immunodeficiency Syndrome | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To provide azithromycin for the treatment of individual patients with proven cryptosporidiosis whose disease has persisted or progressed despite prior therapies.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Cryptosporidiosis infection.
* Life expectancy of at least 1 week.
* Failed or been intolerant to prior therapy with standard antidiarrheal or antibiotic or other therapies for cryptosporidiosis.
* Consent of parent or guardian for patients under the legal age of consent. Patients with documented favorable response to azithromycin under Pfizer protocol 066-143 may receive maintenance therapy under this protocol.

Patients with persistent diarrhea requiring intravenous (IV) fluid therapy to maintain hydration may receive IV azithromycin after approval by the clinical monitor. Patients whose disease worsens despite a minimum of 2 weeks of oral therapy or patients whose disease shows no improvement after 4 weeks of oral therapy will also be considered for a trial period of intravenous azithromycin.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity or significant intolerance to macrolide antibiotics.
* Eligibility and current treatment at a medical center performing study 066-143, another study of azithromycin for treatment of cryptosporidiosis in AIDS patients.

Required:

* Must have failed or been intolerant to prior therapy with standard antidiarrheal or antibiotic therapies for cryptosporidiosis.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Pfizer Central Research, Groton, Connecticut, United States